CLINICAL TRIAL: NCT01709279
Title: Clinical Trial of Autologous Adipose Tissue Derived Stromal Cell Therapy for Ischemic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kanazawa University (Other)
Responsible Party: Principal Investigator, Shuichi Kaneko, Professor, Kanazawa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1133
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Ischemic Heart Failure
Keywords: Ischemic heart failure; Myocardial regeneration; ADRC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adipose tissue derived stromal cells (Other)
  Interventions: Biological: adipose tissue derived stromal cells dosage

INTERVENTIONS:
Biological: adipose tissue derived stromal cells dosage — intra-coronary administration of autologous adipose tissue derived stroma cells

SUMMARY:
Mesenchymal stem cells have capability to differentiate into myocardium, vascular endothelial cell, vascular smooth muscle cell and will be useful for heart regeneration. Adipose tissue is relatively enriched with mesenchymal stem cell compared to bone marrow tissue. In this trial, eligible ischemic heart failure patients will be proceeded intracoronary administration of autologous adipose tissue derived stromal cells by cardiac catheterization.

DETAILED DESCRIPTION:
The population of the ischemic heart failure patients is enormous in Japan and the only radical treatment for them is heart transplantation: however, the number of giving donor is extremely limited. Mesenchymal stem cells have been capable to differentiate into mesodermal-lineage cells as well as endodermal-lineage cells such as myocardial cell. They reside in the mesenchymal tissues such as bone marrows as well as adipose tissues. The latter tissues are relatively enriched with mesenchymal stem cells compared to bone marrow cells. In this study, the ischemic heart failure patients will undergo intracoronary administration of autologous adipose tissue derived stromal cells through cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients occured by prior ischemic event whose ejection fraction must be less than 40%.

Exclusion Criteria:

* Complicated severe other organ disease.
* Patient with malignancy.
* History of chemotherapy or irradiation within 4 weeks.
* Patient with immunodeficiency
* Pregnancy or possibility of pregnancy
* Candidate who are judged to be not applicable to this study by doctors.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
all cause harmful events | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Kanazawa University Hospital, Kanazawa, Ishikawa-ken, Japan